CLINICAL TRIAL: NCT06930612
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of CM512 in Patients With Chronic Rhinosinusitis With Nasal Polyposis
Brief Title: A Study of CM512 in Patients With Chronic Rhinosinusitis With Nasal Polyposis （NEZHA-1）
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM512-102101
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyposis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CM512 Dose 1 (Experimental)
  Interventions: Biological: CM512
- CM512 Dose 2 (Experimental)
  Interventions: Biological: CM512
- CM512 Dose 3 (Experimental)
  Interventions: Biological: CM512
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CM512 — Administered subcutaneous injection
  Arms: CM512 Dose 1; CM512 Dose 2; CM512 Dose 3
Drug: Placebo — Administered subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double blind, placebo-controlled Phase II study to evaluate the efficacy and safety of CM512, and to observe the life quality of subjects, the Pharmacokinetics, Pharmacodynamics and immunogenicity of CM512 in patients with chronic rhinosinusitis with nasal polyposis (CRSwNP).

DETAILED DESCRIPTION:
The study consists of a Screening Period (up to 4 weeks), Treatment Period (24 weeks for double-blind treatment period) and Safety Follow-up Period (12 weeks).

ELIGIBILITY:
Inclusion Criteria:

* with chronic rhinosinusitis with nasal polyposis (CRSwNP).
* Nasal Polyp Score (NPS) of ≥5 with a minimum score of 2 in each nasal cavity.
* Nasal Congestion Score of 2 or 3 at screening period, and at least 2 at baseline.
* Contraception.

Exclusion Criteria:

* Not enough washing out period for previous therapy, e.g., less than 10 weeks or 5 half-lives (whichever is longer) for Interleukin (IL)-4 receptor alpha subunit antagonists, less than 8 weeks or 5 half-lives for biologic therapy/systemic immunosuppressant, less than 6 months for sinus surgery (including polypectomy).With malignant or benign tumor of nasal cavity.
* Vaccination with live attenuated vaccine within 30 days before randomization or during the planned study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-16 (Estimated); Primary Completion 2026-09-16 (Estimated); Study Completion 2026-09-16 (Estimated)

PRIMARY OUTCOMES:
Nasal Polyps Score (NPS) | at week 24
  Change from baseline in the Nasal Polyps Score (NPS) at week 24. NPS score ranges from 0-8 (sum of 0-4 for each nasal passage scores), higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Principal Investigator — Beijing Tong-Ren hospital
Locations (1):
- Beijing Tong-Ren hospital, Beijing, China